CLINICAL TRIAL: NCT05376904
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Parallel-Group, Active-Controlled Study to Evaluate the Efficacy and Safety of Local Administration of HR18034 for Postoperative Analgesia in Subjects Undergoing Hemorrhoidectomy
Brief Title: A Trial of HR18034 for Postoperative Analgesia in Subjects Undergoing Hemorrhoidectomy.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR18034-202
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2022-05

CONDITIONS: Postsurgical Pain Management
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: HR18034 compared with active comparator
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HR18034 dose 1 (Experimental)
  Interventions: Drug: HR18034
- HR18034 dose 2 (Experimental)
  Interventions: Drug: HR18034
- HR18034 dose 3 (Experimental)
  Interventions: Drug: HR18034
- ropivacaine HCl (Active Comparator)
  Interventions: Drug: ropivacaine HCl.

INTERVENTIONS:
Drug: HR18034 — HR18034 low dose
  Arms: HR18034 dose 1
Drug: HR18034 — HR18034 midium dose
  Arms: HR18034 dose 2
Drug: HR18034 — HR18034 high dose
  Arms: HR18034 dose 3
Drug: ropivacaine HCl. — ropivacaine HCl.
  Arms: ropivacaine HCl

SUMMARY:
The study is being conducted to evaluate the efficacy, and safety of HR18034 for postoperative analgesia in subjects undergoing hemorrhoidectomy. To explore the reasonable dosage of HR18034 for postoperative analgesia in subjects undergoing hemorrhoidectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. Subjects requiring hemorrhoidectomy under subarachnoid anesthesia
3. 18 kg/m2 ≤ BMI ≤ 28 kg/m2
4. Conform to the ASA Physical Status Classification
5. Women of childbearing age have a negative pregnancy test and are not nursing

Exclusion Criteria:

1. Subjects with a history of myocardial infarction or unstable angina pectoris
2. Subjects with atrioventricular block or cardiac insufficiency
3. Subjects with a history of ischemic stroke or transient ischemic attack
4. Subjects with a history of mental illness and a history of cognitive impairment epilepsy
5. Subjects with concurrent painful physical condition that may affect postoperative pain assessment
6. Subjects with myelopathy or spinal disease
7. Subjects with a history of hemorrhoidectomy
8. Abnormal values in the laboratory
9. Subject with a history of substance abuse and drug abuse
10. Subject with refractory hypertension
11. History of hypersensitivity or idiosyncratic reactions to amide-type local anesthetics, opioids, or other drugs that may used in study
12. History of substance abuse, drug use and/or alcohol abuse
13. HBsAg, HCVAb, HIV antibody and syphilis antibody tested positive during screening period;
14. Participated in clinical trials of other drugs (received experimental drugs)
15. The inestigators determined that other conditions were inappropriate for participation in this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
AUC of Pain Intensity in rest state | 0~72 hours after administration
  Pain intensity will be evaluated using an 11-point (0-10) Numeric Pain Rating Scale (NPRS), with higher numbers indicating a higher pain intensity, administered over 72 hours.

SECONDARY OUTCOMES:
AUC of Pain Intensity in rest state | 0~24 hours，0~48 hours after administration
  AUC of Pain Intensity in rest state
AUC of Pain Intensity in move state | 0~24 hours，0~48 hours，0~72 hours after administration
  AUC of Pain Intensity in move state
Pain intensity in rest state assessed using an 11-point NPRS ranging | 0~72 hours after administration
  11-point NPRS ranging from a score of 0 to 10
Pain intensity in move state assessed using an 11-point NPRS ranging | 0~72 hours after administration
  11-point NPRS ranging from a score of 0 to 10
Proportion of subjects who doesn't recive rescue analgesic | 0~72 hours after administration
Participant's satisfaction score for analgesia treatment | 72-hours
Investigator's satisfaction score for analgesia treatment | 72-hours

CONTACTS AND LOCATIONS:
Locations (18):
- China (18):
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Tongren Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Dongguan people's Hospital, Dongguan, Guangdong
  - Nanning Second People's Hospital, Nanning, Guangxi
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Traditional Chinese Medicine Hospital of Hebei Province, Shijiazhuang, Hebei
  - Shiyan Taihe Hospital, Shiyan, Hubei
  - the first People's Hospital of Changde, Changde, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Taizhou People's Hospital, Taizhou, Jiangsu
  - Affiliated Zhongshan Hospital of Dalian University, Dalian, Liaoning
  - General Hospital of Northern Theater Command, Shenyang, Liaoning
  - Central Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - the First Affiliated Hospital of Xi'An Jiaotong University, Xi’an, Shanxi
  - The First Affiliated Hospital of Xi'an Medical University, Xi’an, Shanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Jiaxing Second Hospital, Jiaxing, Zhejiang
  - Li Huili Hospital of Ningbo Medical Center, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided